CLINICAL TRIAL: NCT05319379
Title: Clinician Assessment of Patient Dyspnea
Status: Terminated | Type: Observational
Why Stopped: No plans to continue study or publish data.
Sponsor: Rush University Medical Center (Other)
Responsible Party: Principal Investigator, Brady Scott, Associate Professor, Rush University Medical Center
Other Study IDs: 22020104-IRB01
Record Dates: First submitted 2022-03-31; First posted 2022-04-08 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Dyspnea
MeSH Terms: conditions — Dyspnea

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Background: Dyspnea, like pain, is subjective and challenging to assess despite the large number of patients that report shortness of breath. Several studies have shown that physicians and nurses inaccurately assess patient dyspnea. Since respiratory therapists care for many patients at risk for dyspnea, an evaluation of their abilities to evaluate dyspnea is needed. Thus, the plan is to evaluate respiratory therapists' ability to assess a patient's dyspnea level, in addition to nurses and physicians.

Methods: This is a prospective study to evaluate the agreement between dyspnea assessment by a patient and respiratory therapist, nurses, and physicians. The primary aim of this study will be to evaluate clinician ability to assess a patients dyspnea level. The secondary aim of this study is to identify patient characteristics that might influence clinician ability to assess dyspnea.

DETAILED DESCRIPTION:
According to the American Thoracic Society (ATS), the term dyspnea characterizes the subjective experience of breathing discomfort of patients. Dyspnea, like pain, is subjective. Currently, there is no single standard evaluation of dyspnea despite the large number of tools designed to help patients accurately quantify patients who report breathing discomfort.2 Many patients report dyspnea, and studies have shown significant physiological responses associated with breathing discomfort. For example, the amygdala is activated with dyspnea and elicits a sense of impending doom. This is concerning because the prevalence of dyspnea varies widely, from as high as 65% in lung cancer patients to as low as 16% in low-risk population. It appears that the prevalence of dyspnea varies vastly between disease processes, but it not clear if clinicians are able to accurately detect breathing discomfort on routine assessments.

Various efforts have been made to understand how well physicians and nurses assess the dyspnea status of patients. In 2017, Binks et al assessed physicians, nurses, and respiratory therapists on their ability to rate dyspnea in patients requiring mechanical ventilation. The study found that those patients experienced dyspnea and at a significantly higher prevalence than any professional had rated. There was also positive correlation between the amount of discomfort and the degree of underestimation, thus undertreatment which can lead to patient suffering. In a prospective observational study conducted by Puntillo et al, 171 patients considered high risk of dying were assessed for symptoms experienced while in the intensive care unit (ICU). In that study, they found that a significant number of patients had unaddressed symptoms that contributed to unnecessary suffering. Dyspnea was found to be the most distressing symptom that patients experienced. Interestingly, dyspnea was noted in patients that required mechanical ventilation and those that did not.

Stefan et al conducted a study to evaluate the agreement of dyspnea in spontaneously breathing patients with that of the physicians or nurses' assessment. The researchers found that physicians underestimated patients' dyspnea 37.9 % of the time and overestimated 25.8% while nurses underestimated 43.5% and overestimated 12.4%. This is worrisome considering the number of patients that suffer from dyspnea.

Several studies have shown that clinicians responsible for respiratory assessments, like physicians and nurses, often inaccurately assess breathing discomfort. Since respiratory therapists care for many patients at risk for dyspnea, an evaluation of their abilities to assess it should be made. Findings from a study involving respiratory therapists, along with findings from other medical professionals, will provide valuable information for future efforts to better train clinicians on how to best assess dyspnea. The primary aim of this study will be to evaluate clinician (respiratory therapist, nurse, and physician) ability to assess patient dyspnea level. The secondary aims of this study are to identify patient characteristics that might influence clinician ability to assess dyspnea.

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects 18 years and older,
* Admitted to RUMC
* Non-intubated,
* Admitted with a diagnosis of heart failure (HF), chronic obstructive pulmonary disease (COPD), asthma, pneumonia, a generic diagnosis of shortness of breath, or requiring supplemental oxygen support.

Exclusion Criteria:

* Less than 18 years old,
* Non-English-speaking,
* Subjects unable to answer questions about dyspnea for any reason.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients admitted to Rush University Medical Center
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2024-01-03 (Actual); Study Completion 2024-01-03 (Actual)

PRIMARY OUTCOMES:
Agreement between patient and clinician assessment of dyspnea | 1 year

SECONDARY OUTCOMES:
Patient characteristics that might influence clinician ability to assess dyspnea | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States